CLINICAL TRIAL: NCT00376961
Title: A Phase II Study of Combination Rituximab-CHOP and Bortezomib (Velcade®) (R-CHOP-V) Induction Therapy Followed by Bortezomib Maintenance (VM) Therapy for Patients With Newly Diagnosed Mantle Cell Lymphoma
Brief Title: S0601 Rituximab, Combination Chemotherapy, and Bortezomib Followed by Bortezomib Alone in Treating Patients With Newly Diagnosed Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000494646; U10CA032102 (NIH); S0601 (Other: SWOG)
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Results first posted 2013-02-05 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Lymphoma
Keywords: contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Rituximab; Bortezomib; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- R-CHOP + Velcade (Experimental): 6 21-day cycles of standard R-CHOP with 1.3 mg/m^2 Bortezomib given on days 1 and 4 of each cycle. This is followed by 8 3-month cycles of maintenance with 1.3 mg/m^2 Bortezomib on days 1, 4, 8 and 11 of each cycle.
  Interventions: Biological: rituximab; Drug: bortezomib; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate

INTERVENTIONS:
Biological: rituximab — 375 mg/m^2 on day 1 for cycles 1-6.
  Other Names: Rituxan
Drug: bortezomib — 1.3 mg/m^2 on days 1, 4 of cycles 1-6 and on days 1, 4, 8, 11 of cycles 7-14.
  Other Names: Velcade
Drug: cyclophosphamide — 750 mg/m^2 on day 1 of cycles 1-6.
Drug: doxorubicin hydrochloride — 50 mg/m^2 on day 1 of cycles 1-6.
Drug: prednisone — 100 mg on days 1-5 of cycles 1-6.
Drug: vincristine sulfate — 1.4 mg/m^2 on day 1 of cycles 1-6.

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving rituximab together with combination chemotherapy and bortezomib may kill more cancer cells. Giving bortezomib as maintenance therapy may keep the cancer from progressing.

PURPOSE: This phase II trial is studying how well giving rituximab together with combination chemotherapy and bortezomib followed by bortezomib alone works in treating patients with newly diagnosed mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 2-year progression-free survival rate in patients with newly diagnosed mantle cell lymphoma treated with induction therapy comprising rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine, prednisone, and bortezomib followed by bortezomib maintenance (VM) therapy.

Secondary

* Determine the response rate (complete, complete unconfirmed, and partial responses) in patients treated with this regimen.
* Determine the toxicity of VM in these patients.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive R-CHOP-V induction therapy comprising rituximab IV over ≤ 6 hours, cyclophosphamide IV over 15-45 minutes, doxorubicin hydrochloride IV over 5-20 minutes, and vincristine IV over 5-15 minutes on day 1; oral prednisone once daily on days 1-5; and bortezomib IV over 30-90 minutes on days 1 and 4. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. After completion of 6 courses, patients with stable disease or better proceed to bortezomib maintenance therapy.
* Maintenance therapy: Beginning 3 months after completion of R-CHOP-V induction therapy, patients receive bortezomib IV on days 1, 4, 8, and 11. Treatment repeats every 3 months for up to 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 4 years and then annually for 3 years.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed mantle cell lymphoma (MCL) meeting the following criteria:

  * Stage III-IV or bulky stage II disease
  * Confirmation of positivity for the following phenotypes by immunohistochemistry or flow cytometry:

    * Cluster of differentiation antigen 19 (CD19) (or CD20)
    * Cyclin D1 OR evidence of t(11;14) translocation by cytogenetic analysis or fluorescent in situ hybridization
* Newly diagnosed, previously untreated disease
* Bidimensionally measurable disease by conventional techniques

  * No nonmeasurable disease only
* Adequate tumor tissue from original diagnostic specimen available

  * Tissue obtained by needle aspiration or cytology not allowed
* No clinical evidence of central nervous system (CNS) involvement by lymphoma
* Co-registration on protocols SWOG-8947 and SWOG-8819 is strongly encouraged

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No peripheral neuropathy ≥ grade 2
* No hypersensitivity to bortezomib, boron, or mannitol
* No other prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer for which the patient is currently in complete remission, or any other cancer for which the patient has been disease free for the past 5 years
* HIV negative

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, radiotherapy, or antibody therapy for lymphoma
* More than 14 days since prior investigational drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2006-08; Primary Completion 2012-12 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H. Bernstein, MD, Study Chair — James P. Wilmot Cancer Center; Richard I. Fisher, MD, Study Chair — James P. Wilmot Cancer Center
Locations (147):
- United States (147):
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Providence Cancer Center, Anchorage, Alaska
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - North Bay Cancer Center, Fairfield, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Boston University Cancer Research Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Adirondack Cancer Care - Glens Falls, Glens Falls, New York
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - AnMed Cancer Center, Anderson, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - CCOP - Scott and White Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab-CHOP-Bortezomib (R-CHOP-V) Induction: Rituximab-CHOP-Bortezomib (R-CHOP-V) induction is administered every 21 days for 6 cycles (1 cycle = 21 days)
- Bortezomib Maintenance (VM): Bortezomib maintenance (VM) therapy is given 3 months after the completion of R-CHOP-V induction therapy. Treatment with VM is administered once every 3 month for 8 cycles, Cycle 7-14 ( 1 cycle = 3 months)
Period: Initial Registration
Arm/Group | Rituximab-CHOP-Bortezomib (R-CHOP-V) Induction | Bortezomib Maintenance (VM)
Started | 68 | 0
Eligible | 65 | 0
Completed | 61 | 0
Not Completed | 7 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Refusal Unrelated to Adverse Event | 2 | 0
Not completed — Progression/relapse | 1 | 0
Not completed — Ineligible | 3 | 0
Period: Maintenance
Arm/Group | Rituximab-CHOP-Bortezomib (R-CHOP-V) Induction | Bortezomib Maintenance (VM)
Started | 0 | 50
Eligible | 0 | 47
Completed | 0 | 27
Not Completed | 0 | 23
Not completed — Adverse Event | 0 | 1
Not completed — Refusal Unrelated to Adverse Event | 0 | 1
Not completed — Progression/relapse | 0 | 18
Not completed — Ineligible | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Rituximab-CHOP-Bortezomib (R-CHOP-V): R-CHOP-V will be administered for 6 cycles (one cycle is defined as a single 21-day course of treatment).
Arm/Group | Rituximab-CHOP-Bortezomib (R-CHOP-V)
Number analyzed (Participants) | 65
Age, Continuous [Median (Full Range); unit: years] | 61 [36.5 to 85.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 61
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Secondary Outcome: Response Rate in Patients Treated With Rituximab-CHOPbortezomib Induction Therapy (R-CHOP-V) Followed by Bortezomib Maintenance Therapy(VM).
Description: Complete Response(CR) is a complete disappearance of all disease with the exception of nodes. No new lesions. previously enlarged organs must have regressed and not be palpable. Bone marrow(BM) must be negative if positive at baseline. Normalization of markers. CR Unconfirmed (CRU) does not qualify for CR above, due to a residual nodal mass or an indeterminate BM. Partial Response(PR) is a 50% decrease in the sum of products of greatest diameters (SPD) for up to 6 identified dominant lesions, including spleenic and hepatic nodules from baseline. No new lesions and no increase in the size of liver, spleen or other nodes.
Time Frame: At the time of restaging (between Cycles 6 and 7), every 6 months during Cycles 7-14, and at the end of protocol treatment
Population: All eligible patients who started treatment were included in the analysis.
Measure: Number; unit: participants
Groups:
- R-CHOP-V Followed by VM: Rituximab-CHOP-bortezomib induction therapy (RCHOP-V) followed by Bortezomib maintenance therapy (VM). R-CHOP-V is administered for 6 cycles (1 cycle = 21 days). Bortezomib maintenance (VM) therapy is given 3 months after the completion of R-CHOP-V induction therapy. Treatment with VM is administered once every 3 month for 8 cycles, Cycle 7-14 ( 1 cycle = 3 months)
Arm/Group | R-CHOP-V Followed by VM
Number analyzed (Participants) | 65
participants
  Complete Response | 17
  Partial Response | 16
  Unconfirmed Complete Response | 13
  Unconfirmed Partial Response | 1
  No Response | 4
  Assessment Inadequate | 14

2. Primary Outcome: 2-year Progression-free Survival in Patients Treated With Rituximab-CHOP-bortezomib Induction Therapy (RCHOP-V) Followed by Bortezomib Maintenance Therapy (VM)
Description: Measured from date of registration to date of first observation of relapsed or progressive disease, or death due to any cause.
Time Frame: 0-2 years
Population: All eligible patients who started treatment were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | R-CHOP-V Followed by VM
Number analyzed (Participants) | 65
percentage of participants | 62 [49 to 72]

3. Secondary Outcome: 2-year Overall Survival in Patients Treated With Rituximab-CHOP-bortezomib Induction Therapy (RCHOP-V) Followed by Bortezomib Maintenance Therapy (VM)
Description: Measured from date of registration to date of death due to any cause or last contact
Time Frame: 0-2 years
Population: All eligible patients who started treatment were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- R-CHOP-V Followed by VM: Rituximab-CHOP-bortezomib induction therapy (RCHOP-V) followed by Bortezomib maintenance therapy (VM). R-CHOP-V is administered for 6 cycles (1 cycle = 21 dyas). Bortezomib maintenance (VM) therapy is given 3 months after the completion of R-CHOP-V induction therapy. Treatment with VM is administered once every 3 month for 8 cycles, Cycle 7-14 ( 1 cycle = 3 months)
Arm/Group | R-CHOP-V Followed by VM
Number analyzed (Participants) | 65
percentage of participants | 85 [73 to 91]

4. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: Assessed prior to each cycle (for Cycles 2-6), at restaging (between Cycle 6 and 7), every 3 months ( for Cycle 7-14), and at the end of protocol treatment.
Population: Eligible patients who had received any treatment were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | Rituximab-CHOP-Bortezomib (R-CHOP-V) Induction | Bortezomib Maintenance (VM)
Number analyzed (Participants) | 65 | 47
Participants
  Albumin, serum-low (hypoalbuminemia) | 1 | 0
  Anorexia | 1 | 0
  Calcium, serum-low (hypocalcemia) | 1 | 0
  Constipation | 1 | 0
  Dehydration | 1 | 0
  Diarrhea | 3 | 0
  Dizziness | 1 | 0
  Dyspnea (shortness of breath) | 1 | 1
  Edema: limb | 1 | 0
  Fatigue (asthenia, lethargy, malaise) | 6 | 1
  Febrile neutropenia | 12 | 0
  GGT (gamma-glutamyl transpeptidase) | 1 | 1
  Glucose, serum-high (hyperglycemia) | 3 | 0
  Hemoglobin | 3 | 0
  Hypoxia | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 3 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Oral cav-gums | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Sinus | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Ext ear | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Oral cav | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Sinus | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils -Nerve-peri | 1 | 0
  Infection-Other (Specify) | 1 | 0
  Leukocytes (total WBC) | 26 | 0
  Lymphopenia | 15 | 2
  Mucositis/stomatitis (functional/symp) - Oral cav | 1 | 0
  Muscle weakness, not d/t neuropathy - body/general | 1 | 0
  Nausea | 2 | 0
  Neuropathy: CN V Motor-jaw muscles; Sensory-facial | 1 | 0
  Neuropathy: motor | 2 | 0
  Neuropathy: sensory | 2 | 1
  Neutrophils/granulocytes (ANC/AGC) | 34 | 0
  Pain - Head/headache | 0 | 1
  Phosphate, serum-low (hypophosphatemia) | 1 | 0
  Platelets | 11 | 0
  Pneumonitis/pulmonary infiltrates | 1 | 0
  Potassium, serum-low (hypokalemia) | 2 | 0
  Pruritus/itching | 1 | 0
  Renal failure | 1 | 0
  Syncope (fainting) | 2 | 0
  Thrombosis/embolism (vascular access-related) | 1 | 0
  Thrombosis/thrombus/embolism | 1 | 0
  Uric acid, serum-high (hyperuricemia) | 1 | 0
  Urticaria (hives, welts, wheals) | 0 | 1

ADVERSE EVENTS:
Time Frame: Assessed prior to each cycle (for Cycles 2-6), at restaging (between Cycle 6 and 7), every 3 months ( for Cycle 7-14), and at the end of protocol treatment.
Groups:
- Rituximab-CHOP-Bortezomib (R-CHOP-V) Induction: Rituximab-CHOP-Bortezomib (R-CHOP-V) induction is administered every 21 days for 6 cycles (1 cycle= 21 days)
Arm/Group | Rituximab-CHOP-Bortezomib (R-CHOP-V) Induction | Bortezomib Maintenance (VM)
Serious Adverse Events (participants affected / at risk) | 1/65 | 0/47
Other Adverse Events (participants affected / at risk) | 64/65 | 43/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab-CHOP-Bortezomib (R-CHOP-V) Induction (N=65) | Bortezomib Maintenance (VM) (N=47)
Sudden death (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab-CHOP-Bortezomib (R-CHOP-V) Induction (N=65) | Bortezomib Maintenance (VM) (N=47)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 | 0
Hemoglobin (Blood and lymphatic system disorders) | 47 | 15
Auditory/Ear-Other (Specify) (Ear and labyrinth disorders) | 0 | 3
Vision-blurred vision (Eye disorders) | 9 | 0
Watery eye (epiphora, tearing) (Eye disorders) | 6 | 0
Constipation (Gastrointestinal disorders) | 32 | 8
Diarrhea (Gastrointestinal disorders) | 15 | 7
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 4 | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 12 | 3
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 4 | 0
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 10 | 0
Nausea (Gastrointestinal disorders) | 35 | 9
Pain - Abdomen NOS (Gastrointestinal disorders) | 11 | 5
Vomiting (Gastrointestinal disorders) | 12 | 0
Edema: limb (General disorders) | 13 | 3
Fatigue (asthenia, lethargy, malaise) (General disorders) | 52 | 24
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 7 | 0
Pain-Other (Specify) (General disorders) | 0 | 3
Rigors/chills (General disorders) | 11 | 3
Allergic reaction/hypersensitivity (Immune system disorders) | 6 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 0 | 3
Inf w/normal ANC or Gr 1-2 neutrophils - Sinus (Infections and infestations) | 4 | 3
Inf w/normal ANC or Gr 1-2 neutrophils - Up airway (Infections and infestations) | 0 | 8
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 6 | 3
AST, SGOT (Investigations) | 6 | 0
Alkaline phosphatase (Investigations) | 7 | 3
Bilirubin (hyperbilirubinemia) (Investigations) | 0 | 5
Creatinine (Investigations) | 8 | 7
Leukocytes (total WBC) (Investigations) | 45 | 15
Lymphopenia (Investigations) | 27 | 12
Metabolic/Laboratory-Other (Specify) (Investigations) | 10 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 40 | 3
Platelets (Investigations) | 27 | 19
Weight gain (Investigations) | 0 | 5
Weight loss (Investigations) | 10 | 0
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 10 | 0
Anorexia (Metabolism and nutrition disorders) | 17 | 5
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 11 | 5
Dehydration (Metabolism and nutrition disorders) | 5 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 29 | 21
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 4 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 6 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 9 | 3
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 5 | 0
Pain - Back (Musculoskeletal and connective tissue disorders) | 6 | 3
Pain - Bone (Musculoskeletal and connective tissue disorders) | 4 | 0
Pain - Joint (Musculoskeletal and connective tissue disorders) | 15 | 11
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 14 | 8
Dizziness (Nervous system disorders) | 9 | 3
Neuropathy: motor (Nervous system disorders) | 4 | 0
Neuropathy: sensory (Nervous system disorders) | 39 | 34
Pain - Head/headache (Nervous system disorders) | 6 | 8
Taste alteration (dysgeusia) (Nervous system disorders) | 14 | 4
Insomnia (Psychiatric disorders) | 18 | 6
Mood alteration - anxiety (Psychiatric disorders) | 6 | 4
Mood alteration - depression (Psychiatric disorders) | 6 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 10 | 4
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 13
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 5
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 38 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 5
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 | 7
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 4
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 7 | 4
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 0 | 3
Flushing (Vascular disorders) | 5 | 0
Hypertension (Vascular disorders) | 4 | 3
Hypotension (Vascular disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less